CLINICAL TRIAL: NCT05281757
Title: Multicenter Post Market Clinical Follow-Up (PMCF) Study on the Safety and Performance of Ennovate® Complex - A Prospective Study on Scoliosis Patients
Brief Title: Post-Market Clinical Follow-Up Study on the Safety and Performance of Ennovate® Complex
Acronym: COSINE
Status: Recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: Raylytic GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-2022
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Hyperkyphosis; Hyperlordosis; Congenital Scoliosis; Neuromuscular Scoliosis; Idiopathic Scoliosis
Keywords: upper-thoracic spine
MeSH Terms: conditions — Kyphosis; Swayback

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ennovate® Complex: All patients who are treated with the Ennovate® Complex system in accordance with indications given in the instructions for use (IFU)
  Interventions: Device: posterior stabilization for the cervical spine

INTERVENTIONS:
Device: posterior stabilization for the cervical spine — The Ennovate® Complex Spinal System is a posterior stabilization for the Complex and upper-thoracic spine. The implants are used for the posterior multisegmental correction and stabilization over all sections of the spine.

SUMMARY:
Multicenter, multinational Post-Market Clinical Follow-Up (PMCF) study on the safety and performance of Ennovate® Complex - A prospective, pure data collection of all Ennovate® scoliosis patients in selected centers (not interventional, multicentric)

DETAILED DESCRIPTION:
This clinical study is one of the Post-Market Clinical Follow-Up (PMCF) measures that enables the manufacturer to monitor the clinical safety and performance of the Ennovate® Complex system.

The study enables a quick, but detailed implant documentation, which is of great interest for the current and future users of the internal fixation system targeted in this study. It includes the relevant outcomes to evaluate safety and efficacy of the implant system for various indications in deformity disorders.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent in the documentation of clinical and radiological results of patients who are minimum 18 years old
* Informed consent in the documentation of clinical and radiological results of patients AND legal representative (parent) for patients who are younger than 18
* Patient's indication according to IFU
* Patient is not pregnant

Exclusion Criteria:

* Patient's clear unability or unwillingness to participate in follow-up examinations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are treated with the Ennovate® Complex system system in accordance with the indications given in the instructions for use: Hyper- / hypokyphosis, Hyper- / hypolordosis, Scoliosis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change of Pain | preoperatively, at 3-4 months postoperatively and at approximately 12 and 24 months postoperatively
  ain will be assessed by the patient using the Visual Analogue Scale (VAS) which state "0" at one end representing "no pain" and "100" at the opposite end representing "maximal / worst pain".

SECONDARY OUTCOMES:
Change of Quality of Life | preoperatively, at 3-4 months postoperatively and at approximately 12 and 24 months postoperatively
  In order to analyze the quality of life of the patients, the most current questionnaire of the Scoliosis Research Society (SRS), the "SRS-30" is used. The SRS-30 demonstrates how spinal conditions impact quality of life and facilitate comparisons of the quality of life before and after surgical intervention. It is widely used in the evaluation of the treatment of idiopathic scoliosis patients. SRS-30 is a patient self administered questionnaire and has a minimum score of 30 and a maximum score of 150 including postsurgery questions. Each question is scored on 1-5 scale. Questions are sorted into different domains and total and mean scores for each domain are calculated. A total score for the entire questionnaire is also calculated.
Change of Every day life | preoperatively, at 3-4 months postoperatively and at approximately 12 and 24 months postoperatively
  Clinical Results measured by Oswestry Disability Index (ODI). ODI contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel, each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. Each question is scored on a scale of 0 (indicating the least amount of disability) to 5 5 (indicating most severe disability). The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Bone Fusion | at final follow-up approximately 24 months after surgery
  After Complex stabilization fusion of the treated segment is aspired in most cases. The fusion status can be determined from radiographs (static or dynamic). Bony fusion can be characterized quantitatively by the fusion rate.
Cumulative number of Side effects | throughout the follow-up up to 24 months postoperatively
  Occurrence of complications potentially associated with the implanted devices can never be fully excluded during spinal surgery. In order to monitor potential complication and to identify so far unknown complications Adverse Events and Serious Adverse Events deemed related to the investigational device are recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mohd Hisam, Prof. Dr., Principal Investigator — Hospital Universiti Kebangsaan Malaysia (HUKM)
Locations (2):
- University Hospital Brno, Brno, Czechia
- Hospital Universiti Kebangsaan Malaysia (HUKM), Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No